CLINICAL TRIAL: NCT04488016
Title: A 2-Part, Phase I, Open-label, Single-Dose, Sequential Randomized Crossover Study of New Acalabrutinib Tablet in Healthy Subjects to Evaluate Relative Bioavailability, Proton Pump Inhibitor (Rabeprazole) Effect, Food Effect and Particle Size Effect
Brief Title: A Study to Evaluate Relative Bioavailability, Proton Pump Inhibitor (PPI) (Rabeprazole) Effect, Food Effect and Particle Size Effect of New Acalabrutinib Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Acerta Pharma, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8220C00018
Record Dates: First submitted 2020-06-23; First posted 2020-07-27 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Bioavailability; B-cell Lymphoid Cancer
Keywords: Bruton tyrosine kinase (BTK) inhibitor; Proton Pump Inhibitor (Rabeprazole) Effect; Food Effect; Particle Size Effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 -Part 1 (Experimental): Subjects will be randomized to one of 4 sequences ABC, BAC, ABD, or BAD. Subjects will receive 100 mg acalabrutinib capsule, fasted state (>10 h) in Treatment A , 100 mg acalabrutinib tablet (Variant 1), fasted state (>10 h) in Treatment B, 100 mg acalabrutinib tablet (Variant 1), fed state in Treatment C, Rabeprazole 20 mg ×1 (fasted) at 2 hours before administration of 100 mg acalabrutinib tablet (Variant 1)* and following prior administration of rabeprazole 20 mg BID (with meals) on Days -3, -2 and -1 in Treatment D.
  Interventions: Drug: Treatment A- Part 1; Drug: Treatment B- Part 1; Drug: Treatment C - Part 1
- Cohort 2- Part 1 (Experimental): Subjects will be randomized to one of 4 sequences ABC, BAC, ABD, or BAD. Subjects will receive 100 mg acalabrutinib capsule, fasted state (>10 h) in Treatment A , 100 mg acalabrutinib tablet (Variant 1), fasted state (>10 h) in Treatment B, 100 mg acalabrutinib tablet (Variant 1), fed state in Treatment C, Rabeprazole 20 mg ×1 (fasted) at 2 hours before administration of 100 mg acalabrutinib tablet (Variant 1)* and following prior administration of rabeprazole 20 mg BID (with meals) on Days -3, -2 and -1 in Treatment D.
  Interventions: Drug: Treatment A- Part 1; Drug: Treatment B- Part 1; Drug: Treatment C - Part 1
- Cohort 3- Part 1 (Experimental): Subjects will be randomized to one of 4 sequences ABC, BAC, ABD, or BAD. Subjects will receive 100 mg acalabrutinib capsule, fasted state (>10 h) in Treatment A , 100 mg acalabrutinib tablet (Variant 1), fasted state (>10 h) in Treatment B, 100 mg acalabrutinib tablet (Variant 1), fed state in Treatment C, Rabeprazole 20 mg ×1 (fasted) at 2 hours before administration of 100 mg acalabrutinib tablet (Variant 1)* and following prior administration of rabeprazole 20 mg BID (with meals) on Days -3, -2 and -1 in Treatment D.
  Interventions: Drug: Treatment A- Part 1; Drug: Treatment B- Part 1; Drug: Treatment C - Part 1; Drug: Treatment D- Part 1
- Cohort 4 - Part 1 (Experimental): Subjects will be randomized to one of 4 sequences: ABC, BAC, ABD, or BAD. Subjects will receive 100 mg acalabrutinib capsule, fasted state (>10 h) in Treatment A , 100 mg acalabrutinib tablet (Variant 1), fasted state (>10 h) in Treatment B, 100 mg acalabrutinib tablet (Variant 1), fed state in Treatment C, Rabeprazole 20 mg ×1 (fasted) at 2 hours before administration of 100 mg acalabrutinib tablet (Variant 1)* and following prior administration of rabeprazole 20 mg BID (with meals) on Days -3, -2 and -1 in Treatment D.
  Interventions: Drug: Treatment A- Part 1; Drug: Treatment B- Part 1; Drug: Treatment C - Part 1; Drug: Treatment D- Part 1
- Cohort 1- Part 2 (Experimental): Subjects will be randomized to one of 2 sequences in a 2×4 crossover: ABCD or BADC. In Part 2, subjects will be receiving 100 mg acalabrutinib tablet (Variant 1), Variant 2, Variant 3, and 100 mg acalabrutinib solution.
  Interventions: Drug: Treatment A-Part 2; Drug: Treatment B - Part 2; Drug: Treatment C - Part 2; Drug: Treatment D - Part 2
- Cohort 2 - Part 2 (Experimental): Subjects will be randomized to one of 2 sequences in a 2×4 crossover: ABCD or BADC.In Part 2, subjects will be receiving 100 mg acalabrutinib tablet (Variant 1), Variant 2, Variant 3, and 100 mg acalabrutinib solution.
  Interventions: Drug: Treatment A-Part 2; Drug: Treatment B - Part 2; Drug: Treatment C - Part 2; Drug: Treatment D - Part 2

INTERVENTIONS:
Drug: Treatment A- Part 1 — Subjects will receive 100 mg acalabrutinib capsule, fasted state;
  Arms: Cohort 1 -Part 1; Cohort 2- Part 1; Cohort 3- Part 1; Cohort 4 - Part 1
Drug: Treatment B- Part 1 — Subjects will receive 100 mg acalabrutinib tablet (Variant 1), fasted state
  Arms: Cohort 1 -Part 1; Cohort 2- Part 1; Cohort 3- Part 1; Cohort 4 - Part 1
Drug: Treatment C - Part 1 — Subjects will receive 100 mg acalabrutinib tablet (Variant 1), fed state
  Arms: Cohort 1 -Part 1; Cohort 2- Part 1; Cohort 3- Part 1; Cohort 4 - Part 1
Drug: Treatment D- Part 1 — Subjects will receive Rabeprazole 20 mg QD (fasted) at 2 hours before administration of 100 mg acalabrutinib tablet (Variant 1) and following prior administration of rabeprazole 20 mg Twice per day (BID) (with meals) on Days -3, -2 and -1.
  Arms: Cohort 3- Part 1; Cohort 4 - Part 1
Drug: Treatment A-Part 2 — Subjects will receive 100 mg acalabrutinib tablet (Variant 1), fasted state
  Arms: Cohort 1- Part 2; Cohort 2 - Part 2
Drug: Treatment B - Part 2 — Subjects will receive 100 mg acalabrutinib tablet (Variant 2), fasted state
  Arms: Cohort 1- Part 2; Cohort 2 - Part 2
Drug: Treatment C - Part 2 — Subjects will receive 100 mg acalabrutinib tablet (Variant 3), fasted state
  Arms: Cohort 1- Part 2; Cohort 2 - Part 2
Drug: Treatment D - Part 2 — Subjects will receive 100 mg acalabrutinib solution, (Variant 4), fasted state
  Arms: Cohort 1- Part 2; Cohort 2 - Part 2

SUMMARY:
This study will be a 2-part, open-label, single-center relative bioavailability, PPI effect, food-effect and particle size effect randomized crossover study of acalabrutinib tablets in healthy subjects (males or females). The study will be divided in 2 study parts; following a review of the safety and Pharmacokinetics (PK) data from Part 1, the study is planned to be continued with Part 2.

DETAILED DESCRIPTION:
The study will be divided in 2 study parts; Part 1 of this study will be an open-label, 3-treatment-period, 4-treatment, single-center relative bioavailability, PPI effect, and food-effect randomized crossover study of a new acalabrutinib tablet in healthy subjects (males or females).

The relative bioavailability part of Study Part 1 is designed to investigate the PK of the acalabrutinib tablet compared with the PK of acalabrutinib capsule, when administered as a single dose with water under the fasted condition (>10 hours). The PPI effect part of Study Part 1 is designed to compare the PK of acalabrutinib tablet with or without coadministration of the PPI rabeprazole. The food-effect part of Study Part 1 is designed to compare the PK of acalabrutinib tablet under fed and fasted conditions. For each subject, a SmartPill will be administered with 120 mL of still water followed immediately by a single oral dose of acalabrutinib tablet (Treatment B, C or D) or acalabrutinib capsule (Treatment A) administered with 120 mL of still water.

Study Part 1 will comprise:

* A screening period of maximum 28 days;
* Three treatment periods during which subjects will be resident from prior to the evening meal the night before dosing with Investigational medicinal product (IMP) (Day -1) until at least 48 hours after dosing; discharged on the morning of Day 3; and
* A Follow-up Visit within 7 to 10 days. There will be a minimum washout period of at least 7 days between each acalabrutinib administration.

A decision to continue with Study Part 2 will be made following a review of the preliminary data for relative bioavailability (acalabrutinib tablet versus acalabrutinib capsule), food effect, PPI effect, and safety observed in Part 1.

Part 2 of this study will be an open-label, 4-treatment-period, 4-treatment, single-center relative bioavailability, randomized crossover study to determine the effect of particle size on the PK of a single dose of acalabrutinib tablet in healthy subjects (males or females).

This relative bioavailability study is designed to investigate the PK of acalabrutinib tablets with various drug substance particle size distributions and the PK of acalabrutinib solution at a single oral dose of 100 mg under the fasted condition (>10 hours).

Study Part 2 will comprise:

* A screening period of maximum 28 days;
* Four treatment periods during which subjects will be resident prior to the evening meal the night before dosing with IMP (Day -1) until at least 48 hours after dosing; discharged on the morning of Day 3; and
* A Follow-up Visit within 7 to 10 days. There will be a minimum washout period of at least 3 days between each acalabrutinib administration.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy adult male or female subjects aged 18 - 55 years with suitable veins for cannulation or repeated venipuncture.
3. Male subject must adhere to the contraception methods.
4. Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of non-childbearing potential, confirmed at screening.
5. Have a Body mass index (BMI) between 18.5 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive at screening.
6. Understands the study procedures in the Informed Consent Form (ICF) and willing and able to comply with the protocol.
7. Willingness and ability to swallow study drugs, including the SmartPill.
8. Willingness to consume a standardized, high- calorie, high-fat FDA breakfast.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Principal Investigator (PI), may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Evidence of ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infections).
4. Any clinically significant illness, medical/surgical procedure, or trauma within 30 days of the first administration of IMP.
5. Any clinically significant abnormalities in clinical chemistry, hematology, coagulation, or urinalysis results, at screening and first admission to the study unit (first treatment period) as judged by the PI, and defined as: (1) Serum Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), alkaline phosphatase (ALP), and serum bilirubin (total and direct)

   > Upper limit of normal (ULN). (2) Hemoglobin < ULN.
6. Any clinically significant abnormal findings in vital signs at screening and first admission to the study unit (first treatment period), as judged by the PI.
7. Any clinically significant abnormalities on 12-lead ECG at screening and first admission to the study unit (first treatment period), as judged by the PI.
8. Any positive result on screening for serum hepatitis B surface antigen, hepatitis B core antibody (anti-HBc), hepatitis C antibody, and HIV antibody.
9. Known or suspected history of drug abuse, as judged by the PI.
10. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 90 days of the first administration of IMP in this study.

    The period of exclusion begins 90 days after the final dose or 30 days after the last visitwhichever is the longest.
11. Plasma donation within 30 days of screening or any blood donation/loss more than 500 mL during the 90 days prior to screening.
12. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to acalabrutinib or rabeprazole.
13. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 90 days prior to screening.
14. Positive screen for drugs of abuse or cotinine at screening or on each admission to the study center or positive screen for alcohol on each admission to the study center.
15. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
16. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life. Hormone replacement therapy will not be allowed.
17. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the PI.
18. Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate) as judged by the PI. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (e.g., >5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the investigational site.
19. Part 1 only: Inability or unwillingness to swallow SmartPill, including:

Subject has any of the following contraindications for the SmartPill:

1. A history of gastric bezoars
2. Swallowing disorders
3. Suspected or known strictures, fistulas or physiological/mechanical GI obstruction
4. History of GI surgery within 90 days of administration
5. Severe dysphagia to food or pills
6. Crohn's disease or diverticulitis
7. Cardiac pacemakers or other implanted electromedical devices 20 Involvement of any AstraZeneca, Acerta Pharma, Parexel or study site employee or their close relatives. 21 Subjects who have previously received acalabrutinib. 22 Judgment by the PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements. 23 Subjects who cannot communicate reliably with the Investigator. 24 Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax)-Acalabrutinib | Day 1 and Day 2
  Part 1: To assess the relative bioavailability of the acalabrutinib tablet compared with acalabrutinib capsules in fasted state.
  Part 2: To assess the impact of drug substance particle size on the bioavailability of acalabrutinib tablets.
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUClast)-Acalabrutinib | Day 1 and Day 2
  Part 1: To assess the relative bioavailability of the acalabrutinib tablet compared with acalabrutinib capsules in fasted state.
  Part 2: To assess the impact of drug substance particle size on the bioavailability of acalabrutinib tablets.
Area under plasma concentration-time curve from time zero to infinity (AUCinf)-Acalabrutinib | Day 1 and Day 2
  Part 1: To assess the relative bioavailability of the acalabrutinib tablet compared with acalabrutinib capsules in fasted state.
  Part 2: To assess the impact of drug substance particle size on the bioavailability of acalabrutinib tablets.

SECONDARY OUTCOMES:
Cmax -ACP-5862 | Day 1 and Day 2
  Part 1: To assess the ACP-5862 PK profile of the acalabrutinib tablet compared with acalabrutinib capsule in fasted state.
  Part 2: To assess the impact of drug substance particle size on the ACP-5862 PK profile of acalabrutinib tablets.
AUClast-ACP-5862 | Day 1 and Day 2
  Part 1: To assess the ACP-5862 PK profile of the acalabrutinib tablet compared with acalabrutinib capsule in fasted state.
  Part 2: To assess the impact of drug substance particle size on the ACP-5862 PK profile of acalabrutinib tablets.
AUCinf-ACP-5862 | Day 1 and Day 2
  Part 1: To assess the ACP-5862 PK profile of the acalabrutinib tablet compared with acalabrutinib capsule in fasted state.
  Part 2: To assess the impact of drug substance particle size on the ACP-5862 PK profile of acalabrutinib tablets.
Area under the plasma concentration-time curve from time zero to 12 hours post-dose (AUC0-12) - Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
AUClast- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
AUCinf- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
Extrapolated area under the curve from tlast to infinity, expressed as percentage of AUCinf (%AUCextrap)- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
Cmax- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
Half-life associated with terminal slope of a semi-logarithmic concentration-time Curve (t½)- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
Time to reach maximum observed concentration (tmax)- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
Terminal elimination rate constant (Kel)- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
Relative bioavailability (Frel)- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F)- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
Apparent volume of distribution during the terminal phase after extravascular Administration (Vz/F)- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
ACP-5862 (metabolite) to acalabrutinib (parent) ratio (M/P) for Cmax- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
ACP-5862 (metabolite) to acalabrutinib (parent) ratio (M/P) for AUClast- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
ACP-5862 (metabolite) to acalabrutinib (parent) ratio (M/P) for AUCinf- Acalabrutinib and ACP-5862 | Day 1 and Day 2
  Part 1: To evaluate the effects of proton pump inhibitor rabeprazole on acalabrutinib and its metabolite (ACP-5862) PK profiles obtained after dosing the acalabrutinib tablet; To evaluate the effect of food on acalabrutinib and its metabolite (ACP-5862) PK obtained after dosing the acalabrutinib tablet.
  Part 2: To compare PK of acalabrutinib tablet versus acalabrutinib oral solution in healthy subjects.
Number of subjects with adverse events | From Screening to follow-up visit (7 to 10 days after last dose)
  Number of subjects reporting at least one event and number of events where appropriate
Number of subjects with abnormal systolic and diastolic blood pressure | At screening (Day -28), Day -1, and Day 2
  Abnormal values in systolic and diastolic blood pressure.
Number of subjects with abnormal pulse rate | At screening (Day -28), Day -1, and Day 2
  Abnormal values in pulse rate.
Number of subjects with abnormal respiratory rate | At screening (Day -28), Day -1, and Day 2
  Abnormal values in respiratory rate.
Number of subjects with abnormal body temperature | At screening (Day -28), Day -1, and Day 2
  Abnormal values of body temperature.
Number of subjects with abnormal electrocardiogram (12-lead ECG) | At screening (Day -28), Day -1, and Day 2
  Prolongation of the QTc interval.
Number of subjects with abnormal physical examination | At screening (Day -28), Day -1, and Day 2
  Abnormal values in physical examination
Number of subjects with abnormal hematology -Cell count | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  To assess white blood cell count and red blood cell count.
Number of subjects with abnormal electrolytes | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  To assess abnormal serum level of sodium and potassium.
Number of subjects with abnormal hemoglobin (Hb) | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  Abnormal values of hemoglobin
Number of subjects with abnormal hematocrit | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  Abnormal values of hematocrit.
Number of subjects with abnormal mean corpuscular volume (MCV) | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  Abnormal values of MCV
Number of subjects with abnormal mean corpuscular hemoglobin (MCH) | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  Abnormal values of MCH
Number of subjects with abnormal mean corpuscular hemoglobin concentration (MCHC) | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  Abnormal values of MCHC
Number of subjects with abnormal clinical chemistry | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  The laboratory variables to be measured are: bilirubin.
Incidence of abnormal urinalysis | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  The laboratory variables to be measured are: protein in urine. Microscopy (if positive for protein): Casts (Cellular, Granular, Hyaline).
Number of subjects with abnormal glucose (fasting) | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  Abnormal values of glucose (fasting)
Number of subjects with abnormal C-reactive protein (CRP) | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  Abnormal values of CRP.
Number of subjects with abnormal blood urea nitrogen (BUN) | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  Abnormal values of BUN
Number of subjects with abnormal thyroid-stimulating hormone (TSH) | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  Abnormal values of TSH
Number of subjects with abnormal T4 | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  Abnormal values of T4
Number of subjects with abnormal hematology- Differential count | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  To assess neutrophils absolute count, lymphocytes absolute count, monocytes absolute count, eosinophils absolute count, basophils absolute count, platelets, and reticulocytes absolute count.
Percentage of subjects with adverse events | From Screening to follow-up visit (7 to 10 days after last dose)
  Percentage of subjects reporting at least one event and number of events where appropriate
Number of subjects with abnormal electrolytes | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  To assess abnormal serum level of calcium.
Number of subjects with abnormal electrolytes | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  To assess abnormal serum level of phosphate.
Number of subjects with abnormal clinical chemistry | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  The laboratory variables to be measured are: alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST).
Number of subjects with abnormal clinical chemistry | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  The laboratory variables to be measured are: creatinine.
Number of subjects with abnormal clinical chemistry | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  The laboratory variables to be measured are: albumin.
Number of subjects with abnormal clinical chemistry | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  The laboratory variables to be measured are: cystatin C.
Number of subjects with abnormal clinical chemistry | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  The laboratory variables to be measured are: gamma glutamyl transpeptidase.
Number of subjects with abnormal clinical chemistry | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  The laboratory variables to be measured are: urea and uric acid.
Incidence of abnormal urinalysis | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  The laboratory variables to be measured are: glucose in urine.
Incidence of abnormal urinalysis | At screening (Day -28), Day-1, Day 1, Day 2, and Follow-up visit (7-10 days after last dose)
  The laboratory variables to be measured are: blood in urine. Microscopy (if positive blood): RBC, WBC.
Taste | Day 1
  The taste of the acalabrutinib oral solution (Treatment D) will be assessed by a taste and smell questionnaire after the administration of the IMP. Subjects will be asked to complete the questionnaire themselves which will rate questions on the taste of the IMP (sweet, salty, sour, bitter, metallic, hot/spicy, overall taste of the medicine) from 0 to 10 (where 0 is extremely bad and 10 is extremely nice).
Smell | Day 1
  The smell of the acalabrutinib oral solution (Treatment D) will be assessed by a taste and smell questionnaire after the administration of the IMP. Subjects will be asked to complete the questionnaire themselves which will rate questions on the smell of the IMP (extremely bad to extremely nice, whether subjects would take it again) of the medicine) from 0 to 10 (where 0 is extremely bad and 10 is extremely nice).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater,, MD, Principal Investigator — PAREXEL Early Phase Clinical Unit Baltimore
Locations (1):
- Research Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No